CLINICAL TRIAL: NCT04758715
Title: Diet and Microbiome Longitudinal Monitoring With Food Intervention
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nebraska Lincoln (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 20117
Record Dates: First submitted 2021-02-08; First posted 2021-02-17 (Actual); Last update posted 2024-10-21 (Actual); Status verified 2024-10

CONDITIONS: Microbiome, Human; Gastrointestinal Tract

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Food provided (Other): Food provided from a commercial meal service provider for a week
  Interventions: Other: Food provided from a commercial meal service provider for a week

INTERVENTIONS:
Other: Food provided from a commercial meal service provider for a week — Meals from a commercial meal service provider provide for a week to participant

SUMMARY:
The main goal of this project is to identify the microbiome components change in abundance in response to food ingested including provided foods.

ELIGIBILITY:
Inclusion Criteria:

* willing to sign consent and have samples collected,
* able to read and speak English,
* participants must be willing to use an electronic food diary and consume study provided foods,
* only individuals able to provide a US address will be included.

Exclusion Criteria:

* Subjects not able to sign consent on their own accord (ie requiring a Legally Authorized Representative [LAR]),
* Current parenteral nutrition,
* Received cancer treatment within past 6 months prior to signing consent,
* Taken antibiotic treatment within the past 1 month prior to signing consent,
* Received oral x-ray contrast within the past 1 month prior to signing consent,
* Received any type of gastrointestinal bowel preparation in the past 1 month prior to signing consent,
* History of organ transplant,
* Shellfish allergy,
* Insect allergy,
* Cacti allergy,
* Carmine allergy,
* Dragon fruit (pitaya) allergy,

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 65 (Estimated)
Dates: Start 2021-02-02 (Actual); Primary Completion 2030-02-28 (Estimated); Study Completion 2030-02-28 (Estimated)

PRIMARY OUTCOMES:
Microbiota variation | Up to 2 weeks
  Ecological statistics will be used to analyze the longitudinal microbiome composition modification

CONTACTS AND LOCATIONS:
Overall Officials: Jacques Izard, PhD, Principal Investigator — Univeristy of Nebraska-Lincoln
Locations (1):
- University of Nebraska - Lincoln, Lincoln, Nebraska, United States

IPD SHARING:
Plan to Share IPD: No